CLINICAL TRIAL: NCT01568554
Title: Clinical Diagnosis of Acute Porphyria
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Texas (Other); University of Alabama at Birmingham (Other); Icahn School of Medicine at Mount Sinai (Other); University of Utah (Other); Carolinas Medical Center (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Rare Diseases Clinical Research Network (Network)
Responsible Party: Sponsor
Other Study IDs: PC7204; 1U54DK083909 (NIH)
Record Dates: First submitted 2012-02-16; First posted 2012-04-02 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Hereditary Coproporphyria (HCP); Acute Intermittent Porphyria (AIP); Variegate Porphyria (VP)
MeSH Terms: conditions — Coproporphyria, Hereditary; Porphyria, Acute Intermittent; Porphyria, Variegate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group 1: Group 1 will include subjects 15 years of age or older who are a first-degree relative (child, sibling, parent, or grandparent) of an individual with genetically proven acute porphyria (AIP, HCP or VP), and have not had any previous genetic testing for porphyria themselves.
- Group 2 (Not Yet Enrolling): Group 2 will consist of subjects 15 years of age or older who have a history of clinical features suggestive of acute porphyria, such as such as abdominal, back or limb pain, recurrent nausea lasting days, reaction to medications, psychiatric history, or sun sensitivity, and an increase in urinary, fecal or serum porphobilinogen (PBG) and/or porphyrins.
- Group 3: Subjects in Group 3 will participate in the "Follow Up Sub-Study." This group will include individuals who have been seen by one of the Porphyria Consortium physicians/investigators for suspicion of porphyria 10 or more years prior to study initiation, but were not given a diagnosis of porphyria at the time of their initial visit.

SUMMARY:
The purpose of this study is to test whether a focused questionnaire and laboratory tests can better define risk factors associated with possible genetic porphyria. The investigators hypothesize that the genetic carrier state of acute porphyria is distinctive enough that the Genetic Carrier Profile the investigators devise through this study will be useful in identifying carriers of genetic porphyria among the large population with undiagnosed abdominal pain.

DETAILED DESCRIPTION:
The porphyrias are a group of genetic diseases caused by disturbances in the formation of heme, an essential component of hemoglobin and other proteins, leading to either acute (neurologic) and/or chronic (cutaneous) symptoms. Acute porphyria is often difficult to diagnose because symptoms may not be specific and, unless the patient is in an active attack, laboratory values typically may not be useful for diagnosing porphyria. The purpose of this study is to test whether a focused questionnaire and laboratory evaluation tool can better define risk factors associated with possible genetic porphyria. The goals of this study are:

* To determine the presence and number of abnormal lab tests and porphyria-like symptoms in adult family members of the first person in a family who has been diagnosed with a disease of acute porphyria, 50% of whom are expected to carry the same genetic defect of the index case.
* To devise a Genetic Carrie Profile that could be used to screen people in whom the diagnosis of porphyria is being considered.
* To test the Profile in patients with symptoms suggestive of HCP and/or urine tests showing some elevation of porphyrins.
* To explain other possible causes of minor increases in porphyrin levels in patients with recurrent abdominal pain who have not been diagnosed with porphyria

ELIGIBILITY:
Group 1 Inclusion Criteria:

* Be 15 years of age or older
* Be a first-degree relative (child, sibling, parent, or grandparent) of an individual with genetically proven acute porphyria (AIP, HCP or VP)
* Not have had any previous genetic testing for acute porphyria

Group 2 Inclusion Criteria:

* Be 15 years of age or older
* Have a history of suggestive clinical features, such as abdominal, back or limb pain, recurrent nausea lasting days, reaction to medications, psychiatric history, or sun sensitivity.
* An increase in urinary, fecal or serum porphobilinogen (PBG) and/or porphyrins

Groups 1 and 2 Exclusion Criteria:

* Have previously had genetic testing for acute porphyria
* Have a history of "alarm" symptoms, such as anemia, unintentional weight loss, signs of GI (gastrointestinal) bleeding, or dysphagia (difficulty in swallowing).

Follow Up Sub-Study (Group 3) Inclusion Criteria:

* Have been seen by one of the Porphyria Consortium physicians/investigators 10 or more years prior to study initiation
* Had a slight increase in porphyrins during the initial visit
* Not given a diagnosis of porphyria at the time of the visit

Follow Up Sub-Study (Group 3) Exclusion Criteria:

* You have been seen by the Porphyria Consortium physician/investigator less than 10 years prior to study initiation.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Group 1:
  Individuals who are first-degree relatives of a patient with one of the acute porphyrias (AIP, HCP, VP). They will complete questionnaires and laboratory tests, including genetic testing for porphyria. The data will be used to develop a clinical profile for the risk factors associated with the genetic carrier state.
  Group 2:
  Subjects who possibly have acute porphyria, but do not have a confirmed diagnosis based on genetic testing. They will serve to test the validity of the clinical index derived from Group 1.
  Group 3:
  Patients who have been seen by one of the Porphyria Consortium physicians/investigators 10 or more years ago, but were not given a diagnosis of porphyria. They will complete a questionnaire to determine whether they received a porphyria diagnosis, or another diagnosis that might explain the initial presentation.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2011-12; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Presence of positive biochemical features by first-line testing in subjects suspected of being a genetic carrier of acute porphyria | Assessed once at baseline visit for all subjects
  All subjects will be assessed for any elevation of quantitative urine porphobilinogen (PBG).
Presence of positive biochemical features by second-line testing in subjects suspected of being a genetic carrier of acute porphyria | Assessed once at baseline visit for all subjects
  All subjects will be assessed for any elevations of fractionated quantitative urine porphyrins.
Presence of positive biochemical features by second-line testing in subjects suspected of being a genetic carrier of acute porphyria | Assessed once at baseline visit for all subjects
  All subjects will be assessed for any elevations and levels of fractionated quantitative fecal porphyrins.
Clinical features suggestive of the acute porphyria carrier state | Assessed once at baseline visit for all subjects
  Through a focused questionnaire, we will determine the typical duration of pain attacks.
Acute porphyria genetic carrier state | Assessed once at baseline visit for all subjects
  All subjects will undergo DNA analysis to detect a mutation in the HMBS, CPOX, or PPOX genes, respectively.
Other possible causes of mildly elevated porphyrins and recurrent pain | Assessed once during a one-time telephone or in-person interview
  Participants in the Follow-up Sub-study section of this protocol will be interviewed concerning other possible causes of mildly elevated porphyins and recurrent pain. These will be patients previously seen by the investigator who were deemed not to have porphyria.
Presence of heavy metals | Assessed once at baseline visit for all subjects
  All subjects will undergo a blood test to screen for the presence of heavy metals as a cause for minor elevations of porphyrin levels.
Validity of Genetic Carrier Profile | The profile will be tested once during the baseline visit for subjects in Group 2.
  The biochemical and clinical features of genetically proven but asymptomatic HCP will be tabulated and compared to subjects who are not genetic carriers. Its accuracy in predicting risk factors for HCP will be tested in subjects in Group 2.

SECONDARY OUTCOMES:
Frequency of disease manifestations in genetically confirmed AIP and HCP | Assessed annually for 5 years
  Subjects who are confirmed to have AIP and HCP will be assessed at annual follow up visits for the presence and frequency of porphyria symptoms.
Prevalence of HCP in a population with elevation of urine coproporphyrin and pain symptoms. | Assessed once enrollment and genetic testing of subjects in Group 2 are complete - after a 1-year recruitment and enrollment period.
  Based on the number of subjects in Group 2 determined by DNA analysis to have HCP, we will approximate the prevalence of HCP in a population with elevations in coproporphyrin and pain symptoms that are undiagnosed.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Wang, M.D., Study Chair — University of California at San Francisco; Karl E. Anderson, M.D., Principal Investigator — University of Texas; Joseph R. Bloomer, M.D., Principal Investigator — University of Alabama at Birmingham; Robert J. Desnick, Ph.D., M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai; James P. Kushner, M.D., Principal Investigator — University of Utah; Herbert L. Bonkovsky, M.D., Principal Investigator — Carolinas Medical Center and HealthCare System
Locations (6):
- United States (6):
  - UAB Porphyria Center, University of Alabama at Birmingham, Birmingham, Alabama
  - UCSF Porphyria Center, University of California at San Francisco, San Francisco, California
  - Mount Sinai Porphyria Comprehensive Diagnostic & Treatment Center, Mount Sinai School of Medicine, New York, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - UTMB Porphyria Center, University of Texas Medical Branch, Galveston, Texas
  - Porphyria Center, University of Utah, Salt Lake City, Utah